CLINICAL TRIAL: NCT05564715
Title: Cognitive Outcomes of Brain Stimulation As a Later-in-Life Treatment
Acronym: COBALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Alzheimer's Research and Care Consortium (Other)
Responsible Party: Principal Investigator, Christian Lobue, ASSISTANT PROFESSOR - Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2022-0799
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment; Dementia; Amnestic Mild Cognitive Impairment - aMCI
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: In Phase 1, there will be two treatment arms (active and sham). All subjects will have the option to complete active stimulation of HD-tDCS. Those assigned to the sham condition group will have the option to return for active treatment in Phase 2. Each HD-tDCS condition is comprised of 10 days of active or sham stimulation targeting the pre-SMA (supplemental motor area)/sACC (subgenual anterior cingulate cortex) followed by neuropsychological testing after completion of the last session.
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects will be informed that sham and active HD-tDCS will be used in the study, but they will be masked to condition in Phase 1. Aside from the PI, other study team members who perform assessments will be masked to HD-tDCS condition. Questionnaires will be completed examining how well the participants and outcomes assessors were blinded in Phase 1. During Phase 2, individuals who were assigned to the sham condition will be unblinded following all assessments as they will be given the option to return for the active condition. Study team members will become unblinded as a result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Phase 1: Active Treatment (Active Comparator): Participants will receive 10 sessions of active stimulation (1 mA anodal HD-tDCS targeting preSMA/dACC for 20 min) across 2 weeks. Word retrieval and other cognitive tasks will be completed at baseline, immediate follow-up after session 10, and a 2-month follow-up
  Interventions: Device: NeuroElectric StarStim
- Phase 1: Sham Treatment (Sham Comparator): Participants will receive 10 sessions of sham stimulation across 2 weeks. Word retrieval and other cognitive tasks will be completed at baseline, immediate follow-up after session 10, and a 2-month follow-up
  Interventions: Device: Sham Treatment
- Phase 2: Active Treatment (Active Comparator): For Phase 2, participants randomized into the sham group will have the opportunity to return after 2 months from completing Phase 1. They will receive the active treatment while being unblinded to their treatment condition. Following 10 active treatment sessions, word retrieval and other cognitive tasks will again be completed immediately following the last HD-tDCS session and then a 2-month follow-up.
  Interventions: Device: NeuroElectric StarStim

INTERVENTIONS:
Device: NeuroElectric StarStim — 10 sessions of active stimulation (1 mA anodal HD-tDCS targeting preSMA/dACC for 20 min) across 2 weeks
  Other Names: Phase 1/2 Active
  Arms: Phase 1: Active Treatment; Phase 2: Active Treatment
Device: Sham Treatment — Sham stimulation for 10 sessions over 2 weeks
  Arms: Phase 1: Sham Treatment

SUMMARY:
This is a pilot study being done to attempt to improve episodic memory problems in persons with mild cognitive impairment (MCI) or dementia. The pre-supplemental motor area (preSMA) and dorsal anterior cingulate cortex (dACC) have been shown to play a role in episodic memory and language retrieval. Prior studies have suggested that neurostimulation targeting this region can improve episodic memory and word recall. The purpose of this study is to examine the efficacy of high-definition transcranial direct current stimulation (HD-tDCS) to the preSMA/dACC region and its influence on word retrieval and other cognitive functions in patients with MCI or dementia. Entraining the preSMA/dACC circuit with 10 sessions of HD-tDCS will allow us to study whether neurostimulation may be an effective treatment.

DETAILED DESCRIPTION:
The research objective of this study is to examine the efficacy of HD-tDCS to the preSMa/DaCC region and its influence on word retrieval and other cognitive functions in patients with MCI or dementia after 10 sessions of HD-tDCS. There will be two treatment arms: active HD-tDCS (1 mA) and a sham group. For Phase 1, participants will receive 10 sessions of active stimulation (1 mA anodal HD-tDCS targeting preSMA/dACC for 20 min) or sham across 2 weeks. Word retrieval and other cognitive tasks will be completed at baseline, immediate follow-up after session 10, and a 2-month follow-up. For Phase 2, participants randomized into the sham group will have the opportunity to return after 2 months and receive the active treatment while being unblinded to their treatment condition. Following 10 active treatment sessions, word retrieval and other cognitive tasks will again be completed immediately following the last HD-tDCS session and then a 2-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Active diagnosis of mild cognitive impairment or dementia, Female and male subjects, All races/ethnicities, Age 55 years and older, Fluent in English,

Exclusion Criteria:

Lifetime history of major neurologic syndromes (e.g., epilepsy, brain tumor, etc), Substance use disorder within the past year, Has metal fragments in skull/head, Current vision or hearing impairment that interferes with testing, Current medication use known to alter HD-tDCS reactivity

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Changes in Rey Auditory Verbal Learning Test Score | Pre-treatment, post-treatment (an average of 2 weeks), and 8 weeks post-treatment
  The RAVLT is a verbal episodic memory test that is sensitive to mesial and lateral verbal episodic memory circuit dysfunction. The primary outcome measure for this task is the total number of items immediately recalled during the learning trials and after the 20 minute delayed recall trial. Changes in scores from baseline to testing immediately following the completion of the condition will be examined as well as from baseline to 8 months post-treatment.
  RAVLT : Rey Auditory Verbal Learning Test, 0-15 score for each trial, higher scores reflect better performance

SECONDARY OUTCOMES:
Changes in Delis Kaplan Executive Function System (DKEFS) Verbal Fluency Test | Pre-treatment, post-treatment (an average of 2 weeks), and 8 weeks post-treatment
  The DKEFS Verbal Fluency Test is a measure of word retrieval. The task has 3 conditions each lasting 60 seconds, requiring the subject to name words by phonemes, semantic categories, and then switching between two semantic categories. The outcome measure for this task is the total words named for each of the 3 conditions. Changes in scores from baseline to testing immediately following the completion of each condition will be examined as well as from baseline to 8 months post-treatment.
  DKEFS: Delis-Kaplan Executive Function System Verbal Fluency Test, 0-no upper limit for each trial, higher scores reflect better performance
Changes in Boston Naming Test Short Form | Pre-treatment, post-treatment (an average of 2 weeks), and 8 weeks post-treatment
  The Boston Naming Test Short Form has 30 pictures of common objects that upon seeing each picture, individuals need to name the object as soon as one can. The outcome measure for this task is the number of correctly named items. Changes in scores from baseline to testing immediately following the completion of condition will be examined as well as from baseline to 8 months post-treatment.
  BNT: Boston Naming Test - Short Form, 0-30 score, higher scores reflect better performance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No